CLINICAL TRIAL: NCT04570358
Title: Stretching in Children With Spastic Cerebral Palsy
Brief Title: Stretching in Children and Adolescents With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Graz (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Dr. Annika Kruse, Principal investigator, University of Graz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: T1017; T1017-B27 (Other Grant/Funding Number: FWF Austrian Science Fund)
Record Dates: First submitted 2020-09-14; First posted 2020-09-30 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral palsy; Stretching; Muscle-tendon unit; Spasticity; Gait
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Static stretching (Experimental): An 8-week home-based static stretching training for the calf muscles will be performed by group A. Altogether, 10 stretches are performed per leg 4 times a week.
  Interventions: Other: Static stretching
- Control (No Intervention): While group A performs the 8-week static stretching training, group B acts as control group performing its daily life activities as usual.
- Proprioceptive neuromuscular facilitation stretching (Experimental): After group A has finished the 8-week static stretching training, group B starts with the 8-week home-based proprioceptive neuromuscular facilitation stretching training. Altogether, 10 stretches are performed per leg 4 times a week.
  Interventions: Other: Proprioceptive neuromuscular facilitation stretching
- Follow-up (No Intervention): While group B performs the 8-week proprioceptive neuromuscular facilitation stretching, group A is in its follow-up period performing its daily life activities as usual.

INTERVENTIONS:
Other: Static stretching — During the static stretching training for the calf muscles, the ankle joint is moved into maximal dorsiflexion until the point of discomfort is reached. The ankle joint is then held in this maximal position for 30 s followed by a rest period of 30 s. Afterwards, the procedure is repeated with the knee in flexed position to stretch the soleus muscle.
  Arms: Static stretching
Other: Proprioceptive neuromuscular facilitation stretching — During the proprioceptive neuromuscular facilitation stretching, the ankle joint is moved into maximal dorsiflexion. While the foot is kept in this position, the child will perform a (sub-) maximal isometric contraction of the plantar flexors against the resistance of their parents. Afterwards, the ankle joint will be moved further into greater dorsiflexion and is held there for the remaining seconds followed by 30 s of rest. Subsequently, the stretch will be applied with the knee flexed.
  Other Names: PNF
  Arms: Proprioceptive neuromuscular facilitation stretching

SUMMARY:
The primary aim of this study is to gain knowledge about both the effects of a single bout of static and proprioceptive neuromuscular facilitation (PNF) stretching and the effects of 8-week static and PNF stretching training on the calf muscle-tendon properties in children with spastic cerebral palsy (SCP). Furthermore, the effects on joint and muscle function, stretch reflexes, gait, and self-reported gait function and functional performance are examined to receive a comprehensive picture of potential changes.

Further aims of this study are to identify which stretching technique might be more efficient by comparing the effects of both stretching interventions, and to gain information about the influence of foot flexibility on the stretch achieved by the spastic gastrocnemius muscle.

DETAILED DESCRIPTION:
Background: Spastic cerebral palsy (SCP) is a non-progressive neuro-muscular disorder in children resulting from an injury in the central nervous system. Individuals with SCP present with impairments such as hyperreflexia, demonstrate impaired motor control and muscle growth. Manual stretching is an important approach in the physical therapy of individuals with SCP used to increase muscle extensibility and length, decrease muscle stiffness, and to improve functional abilities. However, there are only a few studies that have examined its acute and long-term effects in children with SCP and it is still not clear, if it may lead to the expected changes, and which method might be the most-effective one. Besides static stretching, proprioceptive neuromuscular facilitation (PNF) stretching has been used to aid the rehabilitation of, for example, stroke patients by either facilitating muscle elongation and/or improving muscle strength. Positive effects were found (e.g., increased dorsiflexion, improved gait function, altered tendon properties), which are also clinically relevant for individuals with SCP. However, there is no information about the impact of PNF in this population.

Aims: The primary aim of this study is to gain knowledge about both the effects of a single bout of static and PNF stretching and the effects of 8-week static and PNF stretching training on the calf muscle-tendon properties in children with SCP. Furthermore, the effects on joint and muscle function, stretch reflexes, gait, and self-reported gait function and functional performance are examined to receive a comprehensive picture of potential changes. Further aims of this study are to identify which stretching technique might be more efficient by comparing the effects of both stretching interventions, and to gain information about the influence of foot flexibility on the stretch achieved by the spastic gastrocnemius muscle-tendon unit.

Methods: A randomized controlled trial with a cross-over design will be performed. Prior to the measurements, a familiarization session takes place and both groups will further be examined in three separate measurement sessions. Based on a power calculation and in order to account for possible dropouts, 30 individuals with SCP (age range: 6 to 15 years) will be recruited. The participants will be randomly allocated to either the static stretching or PNF stretching intervention after the familiarization session. Passive muscle-tendon morphological properties will be examined. A manually controlled instrumented spasticity assessment will be performed to test for differences in the reflex responses. Information about the lengthening behavior of the tissues throughout the dorsiflexion rotations will also be collected by use of ultrasound. Isometric muscle strength and the active torque-angle relationship will be investigated using an isokinetic dynamometer. To assess the gait pattern of the children, a gait analysis will be performed by use of an 8-camera motion capture system. In addition, we will examine the participants' gait function and functional performance by use of the Gait Outcomes Assessment List questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* spastic cerebral palsy
* ambulatory children and adolescents
* ability to accept and follow verbal instructions
* no severe contracture of the calf muscles (max. ankle dorsiflexion >= 0°, with knees extended)
* classified as GMFCS level I, II, or III
* aged between 6 and 5 years
* willingness to participate

Exclusion Criteria:

* others than spastic forms of cerebral palsy
* severe mental retardation
* fixed muscle contractures (ankle equinus deformity = max. ankle dorsiflexion <= 0°, with knees extended)
* oral anti-spastic and/or muscle relaxation medication in the last 6 months
* orthopaedic surgery and/or Botulinum toxin type A application in the last 12 months

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Change in mechano-morphological muscle-tendon properties | baseline (T1), post-measurement (T2, 8 weeks), follow-up measurement (T3, 16 weeks)
  Gastrocnemius medialis muscle morphology, muscle stiffness, tendon-aponeurosis length and stiffness, muscle-tendon unit length and stiffness, elongations of the tissues
Change in spasticity/stretch hyperreflexia | baseline (T1), post-measurement (T2, 8 weeks), follow-up measurement (T3, 16 weeks)
  Stretch reflex responses assessed by a manually controlled instrumented spasticity assessment
Change in joint range of motion | baseline (T1), post-measurement (T2, 8 weeks), follow-up measurement (T3, 16 weeks)
  Ankle joint range of motion (maximal plantarflexion - maximal dorsiflexion)
Change in active moment-angle relationship | baseline (T1), post-measurement (T2, 8 weeks), follow-up measurement (T3, 16 weeks)
  Maximum isometric voluntary contractions at specific ankle joint angles (isokinetic dynamometry)

SECONDARY OUTCOMES:
Change in gait characteristics | familiarisation session (T0, 1-week before T1), post-measurement (T2, 8 weeks), follow-up measurement (T3, 16 weeks)
  Gait kinematics of the hip, knee, and ankle joints, gait kinetics (3D motion capture)
Change in self-reported gait, mobility, and functional performance | familiarisation session (T0, 1-week before T1), post-measurement (T2, 8 weeks), follow-up measurement (T3, 16 weeks)
  Gait Outcomes Assessment List (GOAL) questionnaire
Change in maximal isometric muscle strength | baseline (T1), post-measurement (T2, 8 weeks), follow-up measurement (T3, 16 weeks)
  Maximal isometric torque production (isokinetic dynamometry)

OTHER OUTCOMES:
Foot flexibility | familiarisation session (T0, 1 week before baseline assessment)
  Foot flexibility assessment by use of a gonio-dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Annika Kruse, Dr.rer.nat., Principal Investigator — University of Graz, Institute of Human Movement Science, Sport and Health
Locations (1):
- Institute of Human Movement Science, Sport and Health; University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No
It is yet not decided if individual data will be shared with other researchers.

REFERENCES:
- [Background] Lee WY, Park GY, Kwon DR. Comparison of treatment effects between children with spastic cerebral palsy under and over five years after botulinum toxin type a injection. Ann Rehabil Med. 2014 Apr;38(2):200-8. doi: 10.5535/arm.2014.38.2.200. Epub 2014 Apr 29. PMID 24855614
- [Background] Willerslev-Olsen M, Choe Lund M, Lorentzen J, Barber L, Kofoed-Hansen M, Nielsen JB. Impaired muscle growth precedes development of increased stiffness of the triceps surae musculotendinous unit in children with cerebral palsy. Dev Med Child Neurol. 2018 Jul;60(7):672-679. doi: 10.1111/dmcn.13729. Epub 2018 Mar 24. PMID 29573407
- [Background] Barber L, Barrett R, Lichtwark G. Medial gastrocnemius muscle fascicle active torque-length and Achilles tendon properties in young adults with spastic cerebral palsy. J Biomech. 2012 Oct 11;45(15):2526-30. doi: 10.1016/j.jbiomech.2012.07.018. Epub 2012 Aug 3. PMID 22867763
- [Background] Wiart L, Darrah J, Kembhavi G. Stretching with children with cerebral palsy: what do we know and where are we going? Pediatr Phys Ther. 2008 Summer;20(2):173-8. doi: 10.1097/PEP.0b013e3181728a8c. PMID 18480717
- [Background] Sharman MJ, Cresswell AG, Riek S. Proprioceptive neuromuscular facilitation stretching : mechanisms and clinical implications. Sports Med. 2006;36(11):929-39. doi: 10.2165/00007256-200636110-00002. PMID 17052131
- [Background] Zhou Z, Sun Y, Wang N, Gao F, Wei K, Wang Q. Robot-Assisted Rehabilitation of Ankle Plantar Flexors Spasticity: A 3-Month Study with Proprioceptive Neuromuscular Facilitation. Front Neurorobot. 2016 Nov 14;10:16. doi: 10.3389/fnbot.2016.00016. eCollection 2016. PMID 27895574
- [Background] Zhou Z, Zhou Y, Wang N, Gao F, Wang L, Wei K, Wang Q. Changes of Achilles tendon properties via 12-week PNF based robotic rehabilitation of ankle joints with spasticity and/or contracture. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:1214-7. doi: 10.1109/EMBC.2014.6943815. PMID 25570183
- [Derived] Kruse A, Habersack A, Weide G, Jaspers RT, Svehlik M, Tilp M. Eight weeks of proprioceptive neuromuscular facilitation stretching and static stretching do not affect muscle-tendon properties, muscle strength, and joint function in children with spastic cerebral palsy. Clin Biomech (Bristol). 2023 Jul;107:106011. doi: 10.1016/j.clinbiomech.2023.106011. Epub 2023 Jun 7. PMID 37329655